CLINICAL TRIAL: NCT02222376
Title: Effect of Treatment of Diabetic Foot Ulcers With Topic 8% 1-phenyl-5-methyl-2-[1h]-Pyridone (Pirfenidone) Combined With Modified Disulfur Diallyl Oxide (Odd-m) in Gel.
Brief Title: Effect of Topic Pirfenidone in Diabetic Ulcers
Acronym: PirDFI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIA-1031-13/14-1
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic ulcer, diabetic foot
MeSH Terms: conditions — Diabetic Foot | interventions — pirfenidone; Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional treatment (Active Comparator): Weekly ulcer debridement and daily cleansing
  Interventions: Procedure: Debridement
- Pirfenidone (Experimental): Weekly ulcer debridement, daily cleansing, plus twice a day topical pirfenidone application
  Interventions: Drug: Pirfenidone; Procedure: Debridement

INTERVENTIONS:
Drug: Pirfenidone — Twice a day topical application
  Other Names: Kitoscell Q
  Arms: Pirfenidone
Procedure: Debridement — Weekly ulcer debridement

SUMMARY:
Pirfenidone is a synthetic molecule, which acts as a potent modulator of the effect of various cytokines (TNF-α, transforming growth factor-β, platelet derived growth factor and vascular endothelial growth factor, among others) that possesses anti-inflammatory and anti-fibrinolytic properties.

The aim of this study is to compare the effect of topic treatment with pirfenidone compared to conventional treatment in chronic diabetic foot ulcers.

The hypothesis is that treatment with topic pirfenidone in chronic diabetic foot ulcers (Wagner 1 to 2) reduces the ulcer size and shortens the healing time compared to conventional treatment. This is a randomized, controlled and crossover study. Patients will be randomly assigned to conventional treatment or topic pirfenidone for eight weeks. At the end of this period they will change groups. Each week ulcers will be for size, depth, length and evidence of infection. The ulcers will have proper debridement in the conventional treatment group and debridement plus topical pirfenidone application in the pirfenidone group. Subjects will be instructed to do daily ulcer cleansing and for those in the topical pirfenidone group, in addition to cleansing they will be instructed to apply the gel twice a day.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women
2. Type 1 or 2 diabetes
3. Age ≥ 18 years
4. Wagner 1 or 2 diabetic foot ulcer
5. Diabetic ulcer for more than 8 weeks duration
6. Willing to participate in the study with signed informed consent

Exclusion Criteria:

1. Ankle/brachial index < 0.4 (critic ischemia)
2. Use topical or systemic antibiotics
3. Inability to attend to the weekly evaluations
4. Inability to do daily ulcer cleansing
5. Autoimmune diseases
6. Active pharmacologic topical or systemic ulcer treatment
7. Treatment with immunosuppressors such as steroids, radiotherapy, chemotherapy
8. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Ulcer size | 16 weeks

OTHER OUTCOMES:
Healed ulcers | 16 weeks
Adverse effects | 16 weeks
Healing time | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Gomez-Perez, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico